CLINICAL TRIAL: NCT01148199
Title: Self-expandable Metalic Stent Versus Multiple Plastic Stents in Post OLT Biliary Stenosis: Prospective, Randomized, Controlled Trial.
Brief Title: Self-expandable Metallic Stent Versus Multiple Plastic Stents in Post Orthotopic Liver Transplantation Biliary Stenosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, FERNANDA PRATA MARTINS, Attending phisician, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1219-10
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Biliary Anastomotic Stenosis; Biliary Stricture
Keywords: biliary anastomotic stricture; orthotopic liver transplantation; ERCP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple plastic stents (Active Comparator): Multiple plastic stents placement after sphincterotomy and stricutre dilation. ERCP repeated every 3 - 4 months during 1-year
  Interventions: Device: Multiple plastic stents
- Self-expandable metalic stent (Experimental): Self-expandable metalic stent after sphincterotomy. Stent removal scheduled for 6 months
  Interventions: Device: Self-expandable metalic stent

INTERVENTIONS:
Device: Self-expandable metalic stent — Comparison of self-expandable metalic stent versus multiple plastic stents in post OLT biliary stenosis.
  Other Names: Wallflex, Boston Scientific
  Arms: Self-expandable metalic stent
Device: Multiple plastic stents — Comparison of self-expandable metalic stent versus multiple plastic stents in post OLT biliary stenosis.
  Other Names: Boston Scientific; Wilson Cook; Olympus
  Arms: Multiple plastic stents

SUMMARY:
Biliary complications are one of the most common problems after orthotopic liver transplantation (OLT),occurring in up to 24% of patients.

Anastomotic strictures have been endoscopically managed with plastic stents placement. Recently, partially and fully covered metal stents have been alternatively used to treat refractory benign biliary stenosis. The investigators purpose is to compare efficacy and safety of metallic stents versus multiple plastic stents in the endoscopic management of post transplant biliary complications.

DETAILED DESCRIPTION:
Patients with biliary stricture after OLT will be randomly assigned following simple randomization to temporary placement of fully covered self-expandable metal stent (SEMS) or multiple plastic stents placement were randomized according to a computer generated randomization sequence and allocated in a 1:1 ratio to one of two treatment groups.

Final success will be defined as clinical resolution of the stricture without the need to repeat endoscopic, percutaneous or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* post-OLT biliary anastomotic stenosis (at least 1 month post-operative)
* jaundice, cholestasis and/or biliary tree dilation on US

Exclusion Criteria:

* biliary fistulae
* non-anastomotic stricture
* combine anastomotic and non-anastomotic stricture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Post OLT biliary stricture resolution after stent removal | Up to 1 year
  Post OLT biliary stricture resolution will be evaluated during endoscopic stents removal up to 1 year after initial stents placement.

SECONDARY OUTCOMES:
Sustained improvement after endoscopic treatment | 1 year after biliary stenosis resolution
  Stricture resolution persistent after 1 year
Occurence and severity of complications related to the endoscopic procedures | Up to 1 month
  Occurence and severity of complications after therapeutic ERCP will be evaluated and recorded up to 1 month after endoscopic procedures.

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDA P MARTINS, MD, Principal Investigator — Hospital Israelita Albert Einstein; ANGELO P FERRARI, MD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mahajan A, Ho H, Sauer B, Phillips MS, Shami VM, Ellen K, Rehan M, Schmitt TM, Kahaleh M. Temporary placement of fully covered self-expandable metal stents in benign biliary strictures: midterm evaluation (with video). Gastrointest Endosc. 2009 Aug;70(2):303-9. doi: 10.1016/j.gie.2008.11.029. Epub 2009 Jun 11. PMID 19523620
- [Result] Kahaleh M, Behm B, Clarke BW, Brock A, Shami VM, De La Rue SA, Sundaram V, Tokar J, Adams RB, Yeaton P. Temporary placement of covered self-expandable metal stents in benign biliary strictures: a new paradigm? (with video). Gastrointest Endosc. 2008 Mar;67(3):446-54. doi: 10.1016/j.gie.2007.06.057. PMID 18294506
- [Result] Traina M, Tarantino I, Barresi L, Volpes R, Gruttadauria S, Petridis I, Gridelli B. Efficacy and safety of fully covered self-expandable metallic stents in biliary complications after liver transplantation: a preliminary study. Liver Transpl. 2009 Nov;15(11):1493-8. doi: 10.1002/lt.21886. PMID 19877248